CLINICAL TRIAL: NCT03272438
Title: Using a Schedule Intervention to Increase Sustainable Walking Activity in Midlife
Brief Title: Schedule Intervention to Increase Sustainable Walking Activity in Midlife Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Responsible Party: Principal Investigator, Jane Ebert, Associate Professor of Marketing, Brandeis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BrandeisU
Record Dates: First submitted 2017-04-25; First posted 2017-09-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2022-09

CONDITIONS: Physical Activity
Keywords: steps; goals
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three between-subjects conditions: consistent schedule, inconsistent schedule, no schedule. The study is a longitudinal study over 9 weeks, including a baseline week, a 4-week intervention and a follow-up assessment 4 weeks after the intervention.
Who Masked: Participant
Masking Description: Participants are not aware of whether they are in an experimental or control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No schedule control (Active Comparator): This group will receive an accelerometer and daily step goal. They will monitor their steps over the 9 week duration of the study. They will also monitor their steps over the 9 week duration of the study. They will have the same level of contact as the other two conditions.
  Interventions: Device: Accelerometer; Behavioral: Step goal
- Consistent schedule condition (Experimental): This group will receive an accelerometer and daily step goal. They will monitor their steps over the 9 week duration of the study. They will have the same level of contact as the other two conditions. In addition they will plan when, where, and how they will take steps in consistent contexts, i.e., that are very similar from day to day.
  Interventions: Device: Accelerometer; Behavioral: Step goal; Behavioral: Consistent contexts
- Inconsistent schedule condition (Active Comparator): This group will receive an accelerometer and daily step goal. They will monitor their steps over the 9 week duration of the study. They will have the same level of contact as the other two conditions. In addition they will plan when, where, and how they will take steps in inconsistent contexts, i.e., that vary from day to day.
  Interventions: Device: Accelerometer; Behavioral: Step goal; Behavioral: Inconsistent contexts

INTERVENTIONS:
Device: Accelerometer — Participants use an accelerometer to monitor their steps activity
Behavioral: Step goal — Participants are given a daily step goal to aim for
Behavioral: Consistent contexts — Participants plan to take steps in contexts that are similar from day to day
  Arms: Consistent schedule condition
Behavioral: Inconsistent contexts — Participants plan to take steps in contexts that vary from day to day
  Arms: Inconsistent schedule condition

SUMMARY:
While people commonly understand that regular physical exercise conveys many health benefits, only 20% of U.S. adults take regular exercise and they have difficulty maintaining new healthy behaviors. The goal of this study is to use a planning intervention to help establish and maintain a daily step regimen in working midlife adults. The investigators will ask participants to plan when, where, and how to act on a daily walking goal in conjunction with a scheduling intervention to increase the chances that they will maintain this new regimen. The effectiveness of three different scheduling interventions will be compared.

DETAILED DESCRIPTION:
While people commonly understand that regular physical exercise conveys many health benefits, only 20% of U.S. adults take regular exercise and they have difficulty maintaining new healthy behaviors. The goal of this study is to use a planning intervention to help establish and maintain a daily step regimen in working midlife adults. The investigators will ask participants to plan when, where, and how to act on a daily walking goal in conjunction with a scheduling intervention to increase the chances that they will maintain this new regimen. Participants will be randomly assigned to one of three conditions: consistent schedule, inconsistent schedule, no schedule. All participants will be provided with an accelerometer to measure their daily activity and as a behavioral support for our intervention and they will be given a step goal. The goal given to each individual will be to increase immediately their daily steps to a level based on recommended guidelines (e.g., Hill, Wyatt, Reed, and Peters, 2003). The investigators will test which version of the scheduling intervention is most successful for increasing and maintaining step counts. It is predicted that participants in the consistent schedule condition will increase their step count more than those participants in the no schedule control condition, and that they will maintain this activity for a longer period after the intervention period is complete than those participants in the inconsistent schedule condition.

ELIGIBILITY:
Inclusion Criteria:

* currently working 3 or more days (or 24 hours or more) per week;
* physically minimally active (as determined using the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* a recent (within the past 6 months) cardiovascular event, or fall.
* anyone who already exercises regularly, 3 times a week or more for at least 30 minutes, will be excluded

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Physical activity | Daily for 9 weeks
  Number of steps taken each day as measured on accelerometer

SECONDARY OUTCOMES:
Measures of well being | Before and after intervention (5 weeks apart), and at followup (4 weeks later)
  Feelings of satisfaction with life, perceived stress, mood and sleep quality
Physical activity self-efficacy and ease | Weekly for 4 weeks
  Perceived ability and ease of being physically active

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ebert, PhD, Principal Investigator — Brandeis University
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618